CLINICAL TRIAL: NCT00619060
Title: A Phase I Study of Topical Myristyl Nicotinate Cream on Human Skin in Healthy Volunteers
Brief Title: Topical Myristyl Nicotinate Cream on the Skin of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000582627; P30CA023074 (NIH); UARIZ-BIO-07-085 (Other: UA IRB No.)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: skin cancer; healthy, no evidence of disease
MeSH Terms: conditions — Skin Neoplasms | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Myristyl (right), Placebo (Left) (Experimental): Participants apply topical myristyl nicotinate to the right forearm and topical placebo to the left forearm once daily for 4 weeks; Myristyl (Right), Placebo (Left) Topical Myristyl Nicotinate Cream and Placebo
  Interventions: Drug: Topical Myristyl Nicotinate Cream; Drug: Placebo
- Myristyl (Left), Placebo (Right) (Experimental): Participants apply topical myristyl nicotinate to the left forearm and topical placebo to the right forearm once daily for 4 weeks; Myristyl (Left), Placebo (Right)Topical Myristyl Nicotinate Cream and Placebo
  Interventions: Drug: Topical Myristyl Nicotinate Cream; Drug: Placebo

INTERVENTIONS:
Drug: Topical Myristyl Nicotinate Cream — Participants apply topical myristyl nicotinate to one forearm once daily for 4 weeks.
  Other Names: Myristyl; Nicotinate; Cream
Drug: Placebo — Participants apply topical placebo to one forearm once daily for 4 weeks.

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of topical myristyl nicotinate cream may stop skin cancer from forming.

PURPOSE: This randomized phase I trial is studying the side effects and best way to give topical myristyl nicotinate cream on the skin of healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if topical myristyl nicotinate (MN) is a safe, tolerable treatment in healthy volunteers.
* To determine if topically administered MN cream is associated with any significant local or systemic toxicity in normal human subjects in a one-month period.

OUTLINE: Participants are randomized to 1 of 2 treatment arms and serve as their own controls.

* Arm I: Participants apply topical myristyl nicotinate to one forearm and topical placebo to the other forearm once daily for 4 weeks.
* Arm II: Participants receive treatment as in arm I but on opposite forearms. All participants undergo blood collection for chemistry analysis (SMA-20 and CBC) at baseline and at 2 and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older with normal skin
* Have used no topical medications on the skin of the upper extremities, except for emollients or sunscreens, for at least 30 days prior to study entry
* Agree to limit sun exposure as much as possible and wear protective clothing on the forearms in place of using sunscreens or moisturizers
* Ability to understand and willingness to sign an informed consent before initiation of therapy after the nature of the study has been explained to them
* Females must be surgically sterile by hysterectomy or post menopausal

Exclusion Criteria:

* Subjects with no signs of inflammation or irritation of the skin on the forearms
* Subjects with prior history of actinic keratosis or skin cancer on the forearm
* Females of child bearing potential
* Subjects with any concurrent therapy (e.g., retinoids, fluorouracil) on the forearms that may interfere with clinical evaluations
* Subjects taking oral supplemental niacin, by itself or in the form of a multi-vitamin that exceeds 40 mg/day
* No known immunosuppression by virtue of medication or disease, including AIDS patients, subjects taking oral prednisone, and subjects on immunosuppressants/immunomodulators( cyclosporine, chemotherapeutic agents, or biologic therapy), determined by the examining investigator/co-investigator
* Uncontrolled intercurrent illness including, but not limited to any of ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects who have had invasive cancer within the past 5 years
* Skin conditions felt by the study physician to contraindicate enrollment including, but not limited to, psoriasis or atopic dermatitis within a proposed treatment area
* Less than 30 days since prior and no concurrent or planned participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel, MD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Myristyl (Right), Placebo (Left): Participants apply topical myristyl nicotinate to the right forearm and topical placebo to the left forearm once daily for 4 weeks; Myristyl (Right), Placebo (Left)Topical Myristyl Nicotinate Cream and Placebo
  Topical Myristyl Nicotinate Cream and Placebo : Applied topically
Period: Overall Study
Arm/Group | Myristyl (Right), Placebo (Left) | Myristyl (Left), Placebo (Right)
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Myristyl, Placebo: Participants apply topical myristyl nicotinate to the and topical placebo to the other forearm once daily for 4 weeks; Myristyl, Placebo
  Topical Myristyl Nicotinate Cream and Placebo : Applied topically
Arm/Group | Myristyl, Placebo
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events by Treatment.
Description: Comparison of number of participants with adverse events by treatment.
Time Frame: 30 Days
Measure: Number; unit: participants
Groups:
- Myristyl Nicotinate Cream: Participants apply topical myristyl nicotinate to one forearm.
- Topical Placebo Cream: Participants apply topical placebo cream to one forearm.
Arm/Group | Myristyl Nicotinate Cream | Topical Placebo Cream
Number analyzed (Participants) | 22 | 22
participants | 8 | 2
Statistical Analysis 1: Comparison: Myristyl Nicotinate Cream vs Topical Placebo Cream; Test type: Superiority or Other; p = 0.01, Binomial

ADVERSE EVENTS:
Time Frame: 4 weeks; Baseline to completion
Groups:
- Both Forearms: Forearms receiving the Myristyl and Placebo, both arms affected
- Placebo Forearm (Only): Forearms receiving the Placebo
- Myristyl Forearm (Only): Forearms receiving the Myristyl
- Other Non-Derm Events: Systemic Other Adverse Events, i.e. Common Cold, Migraine
Arm/Group | Both Forearms | Placebo Forearm (Only) | Myristyl Forearm (Only) | Other Non-Derm Events
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 1/22 | 2/22 | 8/22 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Both Forearms (N=22) | Placebo Forearm (Only) (N=22) | Myristyl Forearm (Only) (N=22) | Other Non-Derm Events (N=22)
Burning (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Common Cold (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 5 (7) | 0 (0)
Flaking (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (6) | 0 (0)
Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Migraine (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes